CLINICAL TRIAL: NCT03457545
Title: Pilot Study of a Home-based Exercise Intervention to Treat Frailty in Lung Transplant Candidates
Brief Title: Treating Frailty in Lung Transplant Candidates (PREHAB)
Acronym: PREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-17503
Record Dates: First submitted 2018-02-20; First posted 2018-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Advanced Lung Disease

STUDY DESIGN:
Intervention Model Description: Testing a home-based intervention to treat frailty in adult lung transplant candidates using a mobile health technology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Eligible participants will take part in the home-based pulmonary rehabilitation using the Aidcube platform in-person assessment and training with a research coordinator (i.e. physical exercise capacity assessment, SPPB, disability survey, exercise prescription determination, exercise training, dyspnea control techniques) and complete an follow-up assessment at the 8th week.
  Interventions: Behavioral: Home-based pulmonary rehabilitation; Other: Aidcube
- No Intervention (No Intervention): Ineligible participants will receive standard of care

INTERVENTIONS:
Behavioral: Home-based pulmonary rehabilitation — Pilot study of a home-based pulmonary rehabilitation study for lung transplant candidates at the University of California San Francisco
  Arms: Intervention
Other: Aidcube — Participants will be testing and giving feedback on the use of the Aidcube platform in being able to deliver their home-exercise prescription
  Arms: Intervention

SUMMARY:
In this pilot project, 35 lung transplant candidates will be recruited to participate in a three month individualized home-based program focused on exercise and nutrition optimization. This pilot is designed to assess the feasibility of treating frailty before lung transplantation. Participants will complete a 1 day in-person assessment and training session that will include baseline frailty assessment, determination of exercise capacity, and a determination of nutritional status. Based on American Thoracic Society Guidelines and a diet evaluation by a registered dietician, information gathered during the assessment will be used to develop a tailored prescription for exercise and nutrition to be continued at home. Participants will also be taught self-management skills specific to control of dyspnea, fatigue, motivation, and support. Participants will receive training in protocol implementation at home by a coordinator trained in principles of behavior change, adult learning theory, and dyspnea control techniques. Subjects will be provided tablet computers with an app called Aidcube preloaded and taught how to interface with the app. Aidcube is a commercially available exercise platform designed for patients with lung and heart diseases. It was designed with the input of physicians, physical therapists, respiratory therapists, nutritionists who specialize in patients with lung and heart disease and adheres to professional society guidelines for exercise and rehabilitation in patients with lung disease. Subjects will then adhere to a individually tailored home exercise and nutrition program based on their exercise capacity. Aidcube allows clinicians (or in this case the PI and co-PI) the ability to design a customized program of exercises and diet plan through the "provider interface". The subjects interacts with the "patient interface" to complete their exercise program during the 8 week study intervention.

This goal of this pilot project is to determine the feasibility of implementing a home-based exercise and nutrition program with patients with advanced lung disease awaiting lung transplantation.

Information on Aidcube can be found at https://www.aidcube.com.

The overarching aim of this pilot study is preparatory investigation to evaluate the feasibility of performing a home-based intervention to treat frailty in lung transplant candidates.

Specific aims:

* Establish a sampling time frame and recruitment techniques.
* Assess willingness to participate
* Assess adherence and compliance.
* Identify logistical problems in the in-person and at-home components of the intervention
* Determine the resources needed for a full-scale study.
* Provide funding bodies evidence that research team is competent and knowledgeable.
* Provide funding bodies that the study is feasible

DETAILED DESCRIPTION:
Lung transplantation aims to extend survival, reduce disability, and improve health-related quality of life for persons suffering from advanced lung diseases. Despite rigorous candidacy screening practices, improvements in surgical and medical management, and iterative advancements in organ allocation policies, nearly 20% of adults awaiting lung transplantation die or are removed from the waiting list due to disease progression prior to receiving a suitable donor offer1. After lung transplantation, nearly the same proportion of patients dies within the first post-operative year2. Notably, serious morbidity after transplantation is increasing, with resultant disability and associated decrements in health-related quality of life3,4. Although known risk factors for death are already incorporated into lung allocation in the United States (Lung Allocation Score [LAS]), persistently high mortality and increasing morbidity underscore the need to identify novel risk factors for poor outcomes in order to maximize the individual and societal benefit of lung transplantation5.

Frailty- measured by simple, non-invasive clinic based instruments- is an independent risk factor for disability, perioperative complications, and mortality in older medical6-9 and surgical populations10-13. Conceptualized first in the field of geriatrics, frailty is defined as a generalized vulnerability to stressors resulting from an accumulation of physiologic deficits across multiple interrelated systems14. These deficits, in turn, deplete the body's physiologic reserves, resulting in a "state-of-risk" for disproportionate declines in health status following exposure to an additional stressor such as major surgery. Drawing from the geriatrics experience, frailty has become recognized more recently as a risk factor for poor outcomes in solid organ transplantation. Specifically, frailty has been found to be associated with delayed graft function and mortality in kidney transplant recipients and waitlist mortality in liver transplant candidates15-17.

The evaluation of geriatric derived measures is particularly important in contemporary lung transplantation. Indeed, older patients are the fastest growing group of lung transplant candidates in the U.S18. Compared to 8% in 2004, patients aged 65 now account for 30% of annual new recipients, outnumbering those aged 50; those aged 60 account for over half of all new transplants19. This rapid trend has outpaced the evidence base, risk stratification tools, and society guidelines needed to identify which older candidates will do well after lung transplantation. Absent better information, transplant programs have resorted to either ad hoc and admittedly arbitrary chronological age cutoffs or "eyeball tests" of fitness for transplant.

The investigators recently identified frailty as prevalent in lung transplant candidates and independently associated with delisting or death on the waitlist18. Very recently, studies in other populations suggest frailty may be reversible through targeted exercise and nutrition programs. While pulmonary rehabilitation programs may achieve similar goals, a substantial proportion of patients cannot access these programs due to geography or insurance limitations. The investigator's overarching hypothesis is that treating frailty with a home-based intervention before transplant may 1) reduce the risk of death or delisting for becoming too debilitated before transplant and 2) may reduce complications, disability, and possibly mortality after lung transplantation. This proposal seeks to generate critical pilot data needed to inform a larger intervention to treat frailty in lung transplant candidates.

ELIGIBILITY:
Inclusion Criteria:

1. Adult lung transplant candidates in the UCSF Lung Transplant Program aged >=50
2. Ability to understand and speak English or lives with a family member who has the ability to understand and speak English.
3. A diagnosis of chronic obstructive pulmonary disease (COPD) or pulmonary fibrosis (PF).
4. A supplemental oxygen requirement with exercise that can be delivered safely at home using their home oxygen concentrator (as determined by clinically available six-minute walk distance test)
5. Waitilisted or soon to be waitlisted for lung transplantation at UCSF
6. Short Physical Performance Battery (SPBB) frailty score of 9 or less (range 0 - 12; lower scores = worse frailty).
7. Must be an outpatient.
8. Willing and able to come to UCSF Parnassus Campus for 1 day in-person training program.

Exclusion Criteria:

1. Inability to speak or understand English or does not live with a family member who has the abilty to understand and speak English.
2. Subject does not possess home oxygen equipment (if supplemental oxygen is required for exercise)
3. Already or soon to be enrolled in a traditional hospital based pulmonary rehabilitation program
4. Lives alone.
5. A diagnosis of primary or secondary pulmonary hypertension. Diagnosis will be determined by clinically available right heart catheterization pulmonary arterial mean pressure >= 30 mm Hg or transthoracic echocardiogram pulmonary arterial systolic pressure > 50 mm Hg or report of moderate right ventricular dysfunction or worse. These tests are performed as part of routine clinical care in the lung transplant program. Echocardiograms are repeated every 6 months while patients are listed for transplantation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Subject enrollment | Through study completion, an average of 8 to 12 weeks
  Target patients who do not have access to traditional pulmonary rehabilitation programs
Subject attrition | Through study completion, an average of 8 to 12 weeks
  Participant ability to complete program before receiving a lung transplant
Safety | Through study completion, an average of 8 to 12 weeks
  Record number of adverse events, specifically (1) extreme breathlessness, fatigue, and/or weakness, (2) chest pain, (3) severe muscle pain, (4) dizziness or feeling faint, (5) leg pain, weakness or cramping, (6) sweating more than usual, (7) increase in mucus production, and (8) oxygen saturation levels falling below 85% during exercise

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Pre-intervention at week 0 and post-intervention at week 8
  Change in SPPB score (MCID = 1 point)
Six Minute Walk Distance (6MWD) | Pre-intervention at week 0 and post-intervention at week 8
  Change in 6MWD (MCID = 30 meters

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Singer, MD, MS, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valapour M, Skeans MA, Heubner BM, Smith JM, Schnitzler MA, Hertz MI, Edwards LB, Snyder JJ, Israni AK, Kasiske BL. OPTN/SRTR 2012 Annual Data Report: lung. Am J Transplant. 2014 Jan;14 Suppl 1:139-65. doi: 10.1111/ajt.12584. PMID 24373171
- [Background] Yusen RD, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Dobbels F, Goldfarb SB, Levvey BJ, Lund LH, Meiser B, Stehlik J; International Society for Heart and Lung Transplantation. The registry of the International Society for Heart and Lung Transplantation: thirty-first adult lung and heart-lung transplant report--2014; focus theme: retransplantation. J Heart Lung Transplant. 2014 Oct;33(10):1009-24. doi: 10.1016/j.healun.2014.08.004. Epub 2014 Aug 14. No abstract available. PMID 25242125
- [Background] Maxwell BG, Mooney JJ, Lee PH, Levitt JE, Chhatwani L, Nicolls MR, Zamora MR, Valentine V, Weill D, Dhillon GS. Increased resource use in lung transplant admissions in the lung allocation score era. Am J Respir Crit Care Med. 2015 Feb 1;191(3):302-8. doi: 10.1164/rccm.201408-1562OC. PMID 25517213
- [Background] Lyu DM, Zamora MR. Medical complications of lung transplantation. Proc Am Thorac Soc. 2009 Jan 15;6(1):101-7. doi: 10.1513/pats.200808-077GO. PMID 19131535
- [Background] Egan TM, Murray S, Bustami RT, Shearon TH, McCullough KP, Edwards LB, Coke MA, Garrity ER, Sweet SC, Heiney DA, Grover FL. Development of the new lung allocation system in the United States. Am J Transplant. 2006;6(5 Pt 2):1212-27. doi: 10.1111/j.1600-6143.2006.01276.x. PMID 16613597
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Newman AB, Gottdiener JS, Mcburnie MA, Hirsch CH, Kop WJ, Tracy R, Walston JD, Fried LP; Cardiovascular Health Study Research Group. Associations of subclinical cardiovascular disease with frailty. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M158-66. doi: 10.1093/gerona/56.3.m158. PMID 11253157
- [Background] Sancarlo D, Pilotto A, Panza F, Copetti M, Longo MG, D'Ambrosio P, D'Onofrio G, Ferrucci L, Pilotto A. A Multidimensional Prognostic Index (MPI) based on a comprehensive geriatric assessment predicts short- and long-term all-cause mortality in older hospitalized patients with transient ischemic attack. J Neurol. 2012 Apr;259(4):670-8. doi: 10.1007/s00415-011-6241-4. Epub 2011 Sep 23. PMID 21947223
- [Background] Kristjansson SR, Nesbakken A, Jordhoy MS, Skovlund E, Audisio RA, Johannessen HO, Bakka A, Wyller TB. Comprehensive geriatric assessment can predict complications in elderly patients after elective surgery for colorectal cancer: a prospective observational cohort study. Crit Rev Oncol Hematol. 2010 Dec;76(3):208-17. doi: 10.1016/j.critrevonc.2009.11.002. Epub 2009 Dec 14. PMID 20005123
- [Background] Lee DH, Buth KJ, Martin BJ, Yip AM, Hirsch GM. Frail patients are at increased risk for mortality and prolonged institutional care after cardiac surgery. Circulation. 2010 Mar 2;121(8):973-8. doi: 10.1161/CIRCULATIONAHA.108.841437. Epub 2010 Feb 16. PMID 20159833
- [Background] Lee JS, He K, Harbaugh CM, Schaubel DE, Sonnenday CJ, Wang SC, Englesbe MJ, Eliason JL; Michigan Analytic Morphomics Group (MAMG). Frailty, core muscle size, and mortality in patients undergoing open abdominal aortic aneurysm repair. J Vasc Surg. 2011 Apr;53(4):912-7. doi: 10.1016/j.jvs.2010.10.111. Epub 2011 Jan 7. PMID 21215580
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Garonzik-Wang JM, Govindan P, Grinnan JW, Liu M, Ali HM, Chakraborty A, Jain V, Ros RL, James NT, Kucirka LM, Hall EC, Berger JC, Montgomery RA, Desai NM, Dagher NN, Sonnenday CJ, Englesbe MJ, Makary MA, Walston JD, Segev DL. Frailty and delayed graft function in kidney transplant recipients. Arch Surg. 2012 Feb;147(2):190-3. doi: 10.1001/archsurg.2011.1229. PMID 22351919
- [Background] Lai JC, Feng S, Terrault NA, Lizaola B, Hayssen H, Covinsky K. Frailty predicts waitlist mortality in liver transplant candidates. Am J Transplant. 2014 Aug;14(8):1870-9. doi: 10.1111/ajt.12762. Epub 2014 Jun 16. PMID 24935609
- [Background] McAdams-DeMarco MA, Law A, King E, Orandi B, Salter M, Gupta N, Chow E, Alachkar N, Desai N, Varadhan R, Walston J, Segev DL. Frailty and mortality in kidney transplant recipients. Am J Transplant. 2015 Jan;15(1):149-54. doi: 10.1111/ajt.12992. Epub 2014 Oct 30. PMID 25359393
- [Background] Singer JP, Diamond JM, Gries CJ, McDonnough J, Blanc PD, Shah R, Dean MY, Hersh B, Wolters PJ, Tokman S, Arcasoy SM, Ramphal K, Greenland JR, Smith N, Heffernan P, Shah L, Shrestha P, Golden JA, Blumenthal NP, Huang D, Sonett J, Hays S, Oyster M, Katz PP, Robbins H, Brown M, Leard LE, Kukreja J, Bacchetta M, Bush E, D'Ovidio F, Rushefski M, Raza K, Christie JD, Lederer DJ. Frailty Phenotypes, Disability, and Outcomes in Adult Candidates for Lung Transplantation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1325-34. doi: 10.1164/rccm.201506-1150OC. PMID 26258797
- [Background] Chen X, Mao G, Leng SX. Frailty syndrome: an overview. Clin Interv Aging. 2014 Mar 19;9:433-41. doi: 10.2147/CIA.S45300. eCollection 2014. PMID 24672230
- [Background] Cameron ID, Fairhall N, Langron C, Lockwood K, Monaghan N, Aggar C, Sherrington C, Lord SR, Kurrle SE. A multifactorial interdisciplinary intervention reduces frailty in older people: randomized trial. BMC Med. 2013 Mar 11;11:65. doi: 10.1186/1741-7015-11-65. PMID 23497404
- [Background] Fairhall N, Langron C, Sherrington C, Lord SR, Kurrle SE, Lockwood K, Monaghan N, Aggar C, Gill L, Cameron ID. Treating frailty--a practical guide. BMC Med. 2011 Jul 6;9:83. doi: 10.1186/1741-7015-9-83. PMID 21733149
- [Background] Fairhall N, Sherrington C, Lord SR, Kurrle SE, Langron C, Lockwood K, Monaghan N, Aggar C, Cameron ID. Effect of a multifactorial, interdisciplinary intervention on risk factors for falls and fall rate in frail older people: a randomised controlled trial. Age Ageing. 2014 Sep;43(5):616-22. doi: 10.1093/ageing/aft204. Epub 2013 Dec 30. PMID 24381025
- [Background] Latham NK, Harris BA, Bean JF, Heeren T, Goodyear C, Zawacki S, Heislein DM, Mustafa J, Pardasaney P, Giorgetti M, Holt N, Goehring L, Jette AM. Effect of a home-based exercise program on functional recovery following rehabilitation after hip fracture: a randomized clinical trial. JAMA. 2014 Feb 19;311(7):700-8. doi: 10.1001/jama.2014.469. PMID 24549550
- [Background] Roman E, Torrades MT, Nadal MJ, Cardenas G, Nieto JC, Vidal S, Bascunana H, Juarez C, Guarner C, Cordoba J, Soriano G. Randomized pilot study: effects of an exercise programme and leucine supplementation in patients with cirrhosis. Dig Dis Sci. 2014 Aug;59(8):1966-75. doi: 10.1007/s10620-014-3086-6. Epub 2014 Mar 6. PMID 24599772
- See also: Aidcube Website — https://www.aidcube.com

DOCUMENTS (2):
  • Study Protocol (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03457545/Prot_000.pdf
  • Informed Consent Form (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03457545/ICF_001.pdf